CLINICAL TRIAL: NCT00875680
Title: Evaluation of the Efficacy of Autoadjusted Positive Pressure Devices for the Treatment of Obstructive Sleep Apnea Syndrome
Brief Title: Efficacy of autoPPC for the Treatment of Obstructive Sleep Apnea Syndrome (OSAS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Responsible Party: Principal Investigator, Daniel VEALE, Doctor (co-investigator), Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANTADIR CMTS autoPPC 2009
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- autoPPC (Experimental)
  Interventions: Device: autoPPC

INTERVENTIONS:
Device: autoPPC — To test the efficacy of autoPPC machines on residual sleep-related events during a one night autotitration polysomnography.

SUMMARY:
Obstructive Sleep Apnea Syndrome (OSAS) is a common condition that leads to daytime sleepiness and loss of vigilance and, in addition, increased risk of cardiovascular events. The most effective treatment consists in ventilation by mask with continuous positive airway pressure (CPAP), that prevents collapse of the upper airway. However the degree of collapsibility of the pharynx may vary in relation to position, sleep stage, or alcohol or sedative consumption. Thus, CPAP treatment (invented in 1981) has evolved with the development of more sophisticated equipment that permits adapted variations in pressure levels (autoCPAP) with the objective adjusted pressure to avoid airways obstruction with minimal pressure.

Different models of autoCPAP function with different signals and event detection algorithms with different modes of reaction to events. These machines are marketed with CE certification, that guarantees electrical security, but there is to date, no requirement for pre-marketing clinical validation. Nonetheless inadequate treatment may leave patients at risk of accidents and cardiovascular events. These machines can be bench tested using test equipment that can measure with accuracy the response to simulated events, but the testing equipment cannot simulate the diversity of clinical situations, nor the residual level of microarousals that may persist. Thus these bench tests need to be supplemented by clinical studies. The investigators objective is to test the efficacy of these machines on residual sleep-related events during a one night autotitration polysomnography. We develop a prospective, multicentre, non randomised study with autotitration polysomnography only for one night. These clinical results will be compared with the results of bench tests in order to evaluate the pertinence of the bench tests and their eventual utility to simplify clinical evaluation. The perspective of developing a reliable testing protocol may eventually play a role in the certification of these machines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with obstructive sleep apnea syndrome and indication for autoPPC

Exclusion Criteria:

* Patients with COPD, or evolutive heart disease Patients with evolutive cancer Patients already with PPC machine Patients simultaneously included in another clinical study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Residual sleep-related events . | One night of polysomnography

SECONDARY OUTCOMES:
Tolerance and confort of the autoPPC machine | one night

CONTACTS AND LOCATIONS:
Overall Officials: Jean Claude MEURICE, Pr, Principal Investigator — Service explorations fonctionnelles. Hopital La miletrie . POITIERS
Locations (2):
- France (2):
  - MEURICE, Poitiers
  - Service explorations fonctionnelles - Hopital La Miletrie, Poitiers